CLINICAL TRIAL: NCT03343717
Title: Effects of Early Mobilization in Children With Pneumonia
Brief Title: Physiotherapy on Pneumonia in Childrens
Acronym: VAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, DOCTOR, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2.084.580
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Pneumonia
Keywords: Pneumonia, Ventilator-Associated; Mechanical ventilation; Physical therapy
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated | interventions — Rehabilitation; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rehabilitation (Experimental): Phase 1 passive mobilization with 10 repetitions on each joint motion and muscle stretching to the upper.
  Phase 2 - ability to respond to 3 of 5 simple verbal commands. Beginning with passive, active-assisted or active exercises with 5 repetitions in each joint movement in the MMSS and MMII, following the sequence of phase 1.
  Phase 3 - exercises of MMSS with cycle ergometer - 1 series of 1 minute or passive, active-assisted, active or active-resistidos with 5 repetitions in each joint movement, following the sequence of phase 1.
  Interventions: Other: Rehabilitation
- chest physical therapy (Active Comparator): respiratory exercises that include techniques of bronchial hygiene maneuvers with the objective of airway clearance, pulmonary reexpansion techniques for reversal of atelectasis, passive mobilization techniques with the aim of reducing deformities and preserving joint mobility
  Interventions: Other: Chest physical therapy

INTERVENTIONS:
Other: Rehabilitation — physical therapy exercise
  Other Names: physical therapy
  Arms: rehabilitation
Other: Chest physical therapy — chest physical therapy exercise
  Arms: chest physical therapy

SUMMARY:
The children's susceptibility to respiratory problems is due to their anatomical and physiological characteristics; therefore, children with more severe clinical conditions may undergo invasive mechanical ventilation (IMV). However, its prolonged use favors tracheal injury, barotrauma and / or volutrauma, decreased cardiac output and oxygen toxicity, and especially the accumulation of respiratory secretions due to ineffective cough due to non-closure of the glottis and damage in the transport of mucus by the presence of the tracheal tube. Thus, triggering the development of mechanical ventilation-associated pneumonia (VAP), which is defined as a pulmonary infection that arises 48 to 72 hours after endotracheal intubation and the institution of invasive mechanical ventilation. As a consequence, respiratory work is performed by IMV, reducing the work exerted by spontaneous ventilation, causing neuromuscular disorders after 5 to 7 days of IMV, changes in muscle mechanics, reducing the capacity of the diaphragm to generate force, thus contributing to changes in modulation autonomic heart rate, changes in muscular trophism, generating physical deconditioning due to weakness and, finally, an increase in the length of hospitalization and immobilism. From this perspective, early mobilization emerges as a rehabilitation mechanism to improve muscle strength and joint mobility, as well as to improve lung function and respiratory system performance, as well as improved autonomic heart rate modulation. It can facilitate the weaning of IMV, reducing hospitalization time and promoting quality of life after discharge.

DETAILED DESCRIPTION:
We will select 40 volunteers of both sexes and between the ages of 1 and 8 years, with clinical diagnosis of VAP hospitalized in an intensive care unit, which will be submitted, together with the hospital protocol, the protocol of early mobilization. For these patients will be performed physical therapy evaluation in the pre-protocol period, on the second and fourth day of application of the protocol and 1 week at the end of the proposed protocol. For statistical analysis will be compared the pre and post-treatment data found in the evaluations and tabulated in a Microsoft Excel worksheet. BioStat 5.2 software will be used to analyze the results, and the choice of tests for this will depend on the types of distributions found and the homogeneity of the variables.

ELIGIBILITY:
Inclusion Criteria:

* patients on invasive or non-invasive mechanical ventilation for less than 96 hours
* with pneumonia due to invasive mechanical ventilation,
* aged between 1 year and 8 years

Exclusion Criteria:

* Severe Respiratory Failure
* active bleeding
* acute cerebral disorder
* presence of orthopedic contraindications (bone fractures, dislocations, subluxations, postoperative, unstable spine)
* neurological impairment with minimal functionality
* neuromuscular disease

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — 1 year to 8 years
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 5 days
  Influence of exercise on cardiac autonomic modulation

SECONDARY OUTCOMES:
Muscle force | 5 days
  Analysis by Medical Research Council Scale of muscle force. The scale is classified in five grades Grade 5: Muscle contracts normally against full resistance. Grade 4: Muscle strength is reduced but muscle contraction can still move joint against resistance.
  Grade 3: Muscle strength is further reduced such that the joint can be moved only against gravity with the examiner's resistance completely removed. As an example, the elbow can be moved from full extension to full flexion starting with the arm hanging down at the side.
  Grade 2: Muscle can move only if the resistance of gravity is removed. As an example, the elbow can be fully flexed only if the arm is maintained in a horizontal plane.
  Grade 1: Only a trace or flicker of movement is seen or felt in the muscle or fasciculations are observed in the muscle.
  Grade 0: No movement is observed.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Rocha, Doctor, Principal Investigator — Universidade do Estado do Pará
Locations (1):
- Fundação Santa Casa de Misericórdia do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choong K, Koo KK, Clark H, Chu R, Thabane L, Burns KE, Cook DJ, Herridge MS, Meade MO. Early mobilization in critically ill children: a survey of Canadian practice. Crit Care Med. 2013 Jul;41(7):1745-53. doi: 10.1097/CCM.0b013e318287f592. PMID 23507722
- [Result] Choong K, Foster G, Fraser DD, Hutchison JS, Joffe AR, Jouvet PA, Menon K, Pullenayegum E, Ward RE; Canadian Critical Care Trials Group. Acute rehabilitation practices in critically ill children: a multicenter study. Pediatr Crit Care Med. 2014 Jul;15(6):e270-9. doi: 10.1097/PCC.0000000000000160. PMID 24777303
- [Result] Choong K. Early Mobilization in Critically Ill Children: Ready for Implementation? Pediatr Crit Care Med. 2016 Dec;17(12):1194-1195. doi: 10.1097/PCC.0000000000000992. No abstract available. PMID 27918395
- [Derived] Souza GSB, Novais MFM, Lemes GE, de Mello MLFMF, de Sales SCD, Cunha KDC, Rocha LSO, Avila PES, Rocha RSB. Effectiveness of Different Physiotherapy Protocols in Children in the Intensive Care Unit: A Randomized Clinical Trial. Pediatr Phys Ther. 2022 Jan 1;34(1):10-15. doi: 10.1097/PEP.0000000000000848. PMID 34873117